CLINICAL TRIAL: NCT00731874
Title: Thymoglobulin Induction Therapy With Minimal Immunosuppression and Evaluation of Allograft Status by Biopsy and mRNA Profiles (TIMELY Study)
Brief Title: Thymoglobulin Induction Therapy With Minimal Immunosuppression and Evaluation of Allograft Status
Acronym: TIMELY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A higher rate of late rejection was seen in the low tacrolimus arm.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0608008711
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Immunosuppression
Keywords: Kidney transplantation; Immunosuppression; Minimization; Tacrolimus; Prograf; Thymoglobulin
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (6 to 8 ng/mL) (Active Comparator): Target tacrolimus trough concentration of 6 to 8 ng/mL
  Interventions: Drug: Tacrolimus
- Arm 2 (3 to 5 ng.mL) (Active Comparator): Target tacrolimus trough concentration of 3 to 5 ng/mL
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Dosed to achieve target trough concentrations.
  Other Names: Prograf

SUMMARY:
Tacrolimus (Prograf) is a medication that is commonly used in patients who receive a kidney transplant. It is considered to be one of the most important medications that prevent rejection of the transplant kidney by suppressing the immune system. Although tacrolimus is good at preventing rejection, it does have some unwanted side effects. These side effects include high blood pressure, increase in blood sugar, headache, and tremor. In addition, tacrolimus causes some damage to the transplant kidney over time, by causing healthy tissue to turn into scar tissue that does not function as well as healthy tissue. Therefore, kidney function may be reduced over time. In the first three months after kidney transplant, Prograf levels are kept between 8 to 10 ng/mL. This study will compare two groups of patients that will both have their tacrolimus dose reduced slowly over three months to prevent rejection while decreasing the risk of causing toxic effects to the kidney. One group will have their Prograf levels kept between 6 and 8 ng/mL, while the second group will have their levels kept between 3 and 5 ng/mL. We will then compare the two groups to see if there are any differences in their kidney function over time.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety and efficacy of an immunosuppression-minimizing regimen consisting initially of Thymoglobulin induction in combination with tacrolimus, mycophenolate mofetil, and rapid steroid withdrawal. The protocol will minimize long-term calcineurin inhibitor exposure and toxicity by weaning tacrolimus starting at 3 months after transplantation. Patients will be eligible to participate in this study only if they have already consented to participate in another study entitled "The use of urinary PCR test to help detect rejection in kidney transplant patients". In "The use of urinary PCR test to help detect rejection in kidney transplant patients", kidney allograft status (ie. whether or not there is any immunologic activity in the transplant kidney)is characterized with the use of protocol biopsies, diagnostic biopsies, and urinary PCR profiles. At 3 months after transplant, these patients are on an immunosuppression regimen consisting of tacrolimus (Prograf) and mycophenolate mofetil (CellCept). Prograf dosing is managed through the measurement of trough levels. For the first 3 months after transplant, patients are maintained at a trough level between 8 to 10 ng/ml. After 3 months, this target level is lowered in order to minimize long-term exposure to immunosuppressive agents. However, there is no consensus as to what the proper level should be after the first 3 months. Therefore, this study will randomize patients to 2 groups, one group will have their trough level targeted between 6 to 8 ng/mL while the other group will have their trough targeted between 3 and 5 ng/mL. By doing this study, we hope to determine which trough level is best, both for protecting the patient from rejection and protecting the patient from the adverse effects of the immunosuppressive medications.

At New York Weill Cornell Center, we are in a unique position to attempt immunosuppression minimization due to our ability to non-invasively monitor patients using their urine. Previous investigations performed at this center have demonstrated the diagnostic accuracy of mRNA levels of cytotoxic attack molecules in urinary cells. Preliminary data has shown that during acute rejection, Granzyme B and Perforin are strongly expressed in the urine. The sensitivity of the uPCR test was 88% with a specificity of 79%. All kidney transplant recipients at our center are invited to participate in the research study entitled "The use of urinary PCR test to help detect rejection in kidney transplant patients". In this protocol, serial analyses of urinary cells are performed to determine 1) if changes in mRNA levels will predict clinical acute rejection and 2) if these levels correlate with the presence of subclinical acute rejection. Kidney transplant recipients have serial urinary PCR measurements. In addition, patients undergo protocol biopsies of the transplant kidney at 3, 15, and 36 months after transplant. The biopsies help to show the correlation between the PCR results and the pathology of the kidney. It may also serve to detect rejection when the blood tests or urinary PCR do not show it. In a small subset of patients, urinary gene expression profile of cytotoxic attack molecules was able to predict acute rejection prior to clinical diagnosis by renal allograft biopsy.

Because we have the ability to monitor our transplant recipients using the urinary PCR protocol, we can safely minimize tacrolimus exposure over time by monitoring patients non-invasively on a real-time basis. Minimization of immunosuppression over time in a kidney transplant recipient is important in order to prevent or minimize some of the leading causes of kidney graft loss (defined as return to dialysis). Although immunosuppressive medications are excellent at preventing rejection, they do have detrimental effects on the cardiovascular system as well as to the transplant kidney itself. One major cause of kidney graft loss today is chronic allograft nephropathy (CAN). Formerly known as "chronic rejection", CAN has been described as the progressive decline in allograft function that occurs months or years after transplantation, and it is the second leading cause of kidney graft loss. Biopsies of kidney allografts with CAN may show inflammation, fibrosis, glomerulosclerosis, tubular atrophy, and vascular smooth muscle proliferation. The scarring and fibrosis associated with CAN is generally irreversible. A new goal within the modern transplant arena is to prevent CAN from occurring by:

1. decreasing early acute rejection episodes
2. decreasing calcineurin inhibitor-related nephrotoxicity

With the use of modern immunosuppressive agents and induction therapy, we have already decreased early acute rejection episodes significantly. At this time, we now want to begin to study the potentially beneficial effects that calcineurin inhibitor withdrawal may have on kidney function as well as long-term graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Renal allograft recipients who received a steroid-sparing immunosuppression protocol with rabbit anti-thymocyte globulin (Thymoglobulin) induction
* Patient must have previously enrolled in protocol entitled "The use of urinary PCR test to help detect rejection in kidney transplant patients"
* Recipients must agree to undergo all standard post-transplant protocol biopsies
* Recipients must be at least 3 months post-transplant and the three most recent urinary profiles must demonstrate immunologic quiescence as determined by measurement of Granzyme B and Perforin copy numbers
* Patient must provide informed consent to participate in the research study

Exclusion Criteria:

* Patient is a high-risk recipient (defined as peak or current PRA >50% or a re-transplant recipient who lost prior graft within 1 year due to immunologic reasons)
* Patients who require maintenance steroids for another medical condition (such as asthma)
* Patients who are taking less than 1 gram/day of mycophenolate mofetil
* Multiple organ transplant recipients (such as kidney-pancreas)
* Patients with one or more acute rejection episodes within the first 3 months after transplant
* Three-month protocol biopsy showing clinical acute rejection (BANFF grade 1a or higher)
* Patient with documented or suspected non-compliance with transplant medications in the first 3 months after transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Kapur, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College/NewYork-Presbyterian Hospital, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 subjects consented for the study; 11 were enrolled but not randomized due to the following: withdrew consent/refused transplant biopsy (n=4); donor specific antibody detected during screening (n=3); excluded by findings of kidney transplant biopsy (n=2); fluctuation in renal function (n=1); study terminated prior to randomization (n=1).
Groups:
- Arm 1 (Target Tacrolimus 6 to 8 ng/mL): Target tacrolimus trough concentration of 6 to 8 ng/mL
  Tacrolimus: Dosed to achieve target trough concentrations.
- Arm 2 (Target Tacrolimus 3 to 5 ng/mL): Target tacrolimus trough concentration of 3 to 5 ng/mL
  Tacrolimus: Dosed to achieve target trough concentrations.
Period: Overall Study
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Started | 10 | 13
Completed | 10 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL) | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.3) | 56.1 (10.2) | 52.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 11 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy-confirmed Acute Rejection and/or Progression of Histologically Proven Chronic Allograft Nephropathy at 15 Months After Transplantation.
Time Frame: 15 months post-transplant
Measure: Number; unit: participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 10 | 13
participants | 0 | 1

2. Secondary Outcome: Patient Survival
Time Frame: 36 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 10 | 13
Participants | 10 | 13

3. Secondary Outcome: Graft Survival
Time Frame: 36 months post-transplant
Population: Data are not included for one subject because one subject was lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 10 | 12
Participants | 10 | 12

4. Secondary Outcome: Change in Incidence and Severity of Interstitial Fibrosis/Tubular Atrophy (IF/TA) From the Baseline 3-month Biopsy to the 36-month Biopsy
Description: Compared to the baseline biopsy performed at the time of study entry at 3 months, was there new development (incidence) or progression (severity) of interstitial fibrosis/tubular atrophy (formerly called chronic allograft nephropathy) in the biopsy performed at 36 months.
Time Frame: 36 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 10 | 13
Participants
  Progression of IFTA | 2 | 5
  New IFTA | 2 | 1
  Stable Biopsy | 4 | 6
  No Data | 2 | 1

5. Secondary Outcome: Renal Function (Estimated Glomerular Filtration Rate)
Time Frame: 36 months post-transplant
Population: Data are not included for one subject because one subject was lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 10 | 12
Participants
  eGFR>60 | 2 | 5
  eGFR 50-59 | 4 | 3
  eGFR 40-49 | 2 | 1
  eGFR 30-39 | 1 | 2
  eGFR 20-29 | 1 | 1

6. Secondary Outcome: Development of Donor Specific Antibody (DSA)
Description: Percent of subjects who developed new donor specific antibody (mean fluorescence intensity > 3,000) after enrollment, within 36 months of transplant
Time Frame: 36 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 10 | 13
Participants | 0 | 5

7. Secondary Outcome: Incidence of Acute Rejection
Description: Incidence of biopsy-proven acute rejection
Time Frame: 36 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 10 | 13
Participants | 0 | 5

8. Secondary Outcome: Severity of Acute Rejection (by Banff Criteria and Need for Anti-lymphocyte Agents to Treat Acute Rejection)
Description: The severity of acute rejection may be assessed by the Banff criteria. The Banff Classification of Allograft Pathology is an international consensus classification for the reporting of renal allograft biopsies, and provides critical information enabling the diagnosis and grading of pathologic changes, can help to predict response to treatment, and can help to determine the long-term prognosis of the organ. Anti-lymphocyte agents (specifically rabbit anti-thymocyte globulin) are used to treat more severe cases of acute rejection, and thus may serve as a surrogate marker of severity.
Time Frame: 36 months post-transplant
Population: Data reported only for those subjects who developed acute rejection during the study, per protocol. Three of the 5 subjects in Arm 2 with rejection were treated with rabbit anti-thymocyte globulin.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 0 | 5
Participants
  Mixed T cell and Antibody Mediated Rejection | 0 | 3
  Antibody Mediated Rejection | 0 | 2

9. Secondary Outcome: Incidence of Opportunistic Infection
Time Frame: 36 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 10 | 13
Participants | 1 | 1

10. Secondary Outcome: Development of New Onset Diabetes Mellitus
Time Frame: 36 months post-transplant
Population: Only subjects who did not have a diagnosis of diabetes mellitus at transplant are included, per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Number analyzed (Participants) | 8 | 9
Participants | 1 | 2

ADVERSE EVENTS:
Arm/Group | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 3/10 | 7/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Target Tacrolimus 6 to 8 ng/mL) (N=10) | Arm 2 (Target Tacrolimus 3 to 5 ng/mL) (N=13)
Pain, Hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Cytomegalovirus viremia (Infections and infestations) | 0 (0) | 1 (1)
Antibody-mediated rejection (Renal and urinary disorders) | 0 (0) | 5 (5)
Non-melanoma skin cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Strongyloides infection (Infections and infestations) | 1 (1) | 0 (0)
Endometritis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The population reported is small because the study was stopped early due to the increase in late antibody mediated rejection (occurring after month 15) that was seen in Arm 2 (target tacrolimus trough 3 to 5 ng/mL).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No